CLINICAL TRIAL: NCT05286359
Title: Multi-site, Prospective, Clinical Performance Evaluation of NxTekTM Malaria Pf Plus Rapid Diagnostic Test Device and NxTekTM Malaria Pf/Pv Plus Rapid Diagnostic Test (RDT) Device for the Detection of Plasmodium Infections in Patients With Symptoms Suggestive of Malaria
Brief Title: Performance Evaluation of Malaria Plus Rapid Diagnostic Tests (RDTs) for the Detection of Plasmodium Infections in Patients With Symptoms Suggestive of Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDRD-G-001-P
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Malaria
Keywords: Plasmodium infection; Plasmodium falciparum; Plasmodium vivax
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Malaria, Vivax

STUDY DESIGN:
Masking Description: The staff conducting the trial assays will be blinded to any results already available from the investigational, comparator or reference test.
  All RDTs will be read by two blinded operators, with a third operator for discrepant results
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NxTekTM Malaria Plus Rapid Diagnostic Test (RDT) Devices (Experimental)
  Interventions: Diagnostic Test: NxTekTM Malaria Pf Plus Rapid Diagnostic Test Device

INTERVENTIONS:
Diagnostic Test: NxTekTM Malaria Pf Plus Rapid Diagnostic Test Device — NxTekTM Malaria Pf/Pv Plus: A sensitive rapid chromatographic immunoassay for the qualitative detection of histidine-rich protein 2 (HRP2) and Plasmodium lactate dehydrogenase (pLDH) of Plasmodium falciparum(P.f.) on one test line and of pLDH of Plasmodium vivax (P.v.) malaria on a second test line in human whole blood. This test is a lateral flow test for in vitro professional diagnostic use and intended as an aid to early diagnosis of Malaria infection in-patients with clinical symptoms.
  NxTekTM Malaria Pf Plus: A sensitive rapid chromatographic immunoassay for the qualitative detection of histidine-rich protein 2 (HRP2) and pLDH on a single test line of Plasmodium falciparum(P.f.) malaria in human whole blood. This test is a lateral flow test for in vitro professional diagnostic use and intended as an aid to early diagnosis of Malaria infection in-patients with clinical symptoms.
  Other Names: NxTekTM Malaria Pf/Pv Plus Rapid Diagnostic Test Device

SUMMARY:
This trial is part of a portfolio of studies designed to assess the clinical and operational performance of Abbott's NxTekTM Malaria Pf Plus and NxTekTM Malaria Pf/Pv Plus Rapid Test Devices.

DETAILED DESCRIPTION:
A prospective cross-sectional multi-center diagnostic accuracy trial in intended-use settings of the:

1. NxTekTM Malaria Pf/Pv Plus Rapid Test Device for the qualitative detection histidine-rich protein II (HRP-II antigens) and pLDH of Plasmodium falciparum (P.f) and Plasmodium vivax (P.v) malaria in human whole blood.
2. NxTekTM Malaria Pf PlusRapid Test Device for the qualitative detection of histidine-rich protein II (HRP-II antigens) and pLDH of Plasmodium falciparum (P.f) malaria in human whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5years old or older
* Presenting at the trial site with fever or a history of fever (axillary temp ≥ 37.5C) during the preceding 48hours
* Freely agreeing to participate by providing informed consent (and assent, if applicable)

Exclusion Criteria:

* Presence of symptoms and signs of severe illness and/or central nervous system infections as defined by WHO guidelines.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Assess the sensitivity, specificity, positive and negative predicting values (PPV and NPV) [altogether referred to hereafter as "diagnostic accuracy"] of NxTekTM Malaria Pf Plus | 6 months
  To assess the sensitivity, specificity, positive and negative predicting values (PPV and NPV) [altogether referred to hereafter as "diagnostic accuracy"] of NxTekTM Malaria Pf Plus in intended use settings for detecting P.f. infections in capillary whole blood samples collected prospectively from patients with symptoms suggestive of malaria (e.g. febrile).
To assess the diagnostic accuracy of NxTekTM Malaria Pf/Pv Plus. | 6 months
  To assess the diagnostic accuracy of NxTekTM Malaria Pf/Pv Plus in intended use settings for detecting P.f. and P.v. infections in capillary whole blood samples collected prospectively from patients with symptoms suggestive of malaria (e.g. febrile).

SECONDARY OUTCOMES:
Estimates of diagnostic accuracy characteristics with 95% confidence intervals of comparator tests (05FK50, 05FK80, 05FK120, LM) | 6 months
  Estimates of diagnostic accuracy characteristics with 95% confidence intervals of comparator tests (05FK50, 05FK80, 05FK120, LM), using the reference test as standard of truth for the detection of P. falciparum and, when relevant, P.v. infections in patients with symptoms suggestive of malaria
Estimates of diagnostic accuracy characteristics with 95% confidence intervals ofthe index tests for the detection of P.f.infections with hrp2 and/or hrp3 deletions | 6 months
  Estimates of diagnostic accuracy characteristics with 95% confidence intervals of the index tests for the detection of P.f. infections with hrp2 and/or hrp3 deletions in patients with symptoms suggestive of malaria

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lemu Golassa, PhD, Principal Investigator — Addis Ababa University
Locations (1):
- Medical Parasitology Research Unit, Aklilu Lemma Institute of Pathobiology (ALIPB), Addis Ababa University (AAU)., Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mandefro A, Ding XC, Farge J, Alemayehu GS, Tadele G, Mekonen B, Gebrehiwot Y, Berhe N, Erko B, Slater HC, Bizilj GT, Barney R, Golden A, Domingo GJ, Golassa L. Performance of a novel P. falciparum rapid diagnostic test in areas of widespread hrp2/3 gene deletion. Clin Infect Dis. 2025 Apr 24:ciaf212. doi: 10.1093/cid/ciaf212. Online ahead of print. PMID 40274531